CLINICAL TRIAL: NCT05854706
Title: Antidepressant Effect of Prolonged Intermittent Theta-burst Stimulation on Serum Brain-derived Neurotrophic Factor Levels of Patients With Depression: A Randomized, Double-Blind, Sham-Controlled Study
Brief Title: The Effect of Theta-burst Stimulation on Serum BDNF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCHIRB-11003020
Record Dates: First submitted 2023-04-18; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-02

CONDITIONS: Gambling Disorder
Keywords: Brain-Derived Neurotrophic Factor, Theta Burst Stimulation
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Experimental): Prolonged iTBS sessions are scheduled daily in a 5-day sequence for 10 sessions over two weeks
  Interventions: Device: Theta Burst Stimulation
- Sham arm (Sham Comparator): Sham stimulation sessions are scheduled daily in a 5-day sequence for 10 sessions over two weeks
  Interventions: Device: Theta Burst Stimulation

INTERVENTIONS:
Device: Theta Burst Stimulation — Theta Burst Stimulation

SUMMARY:
The goal of this clinical trial is to investigate the effect of theta burst stimulation for depression and serum brain-derived neurotrophic factor (BDNF) in individuals with major depression. The main question it aims to answer is whether 10 sessions of theta burst stimulation can influence the serum level of BDNF.

Participants will be randomized into active group and sham group. Researchers will compare the level of BDNF in these groups.

DETAILED DESCRIPTION:
There is an increasing evidence that the BDNF could be involved in the mode of action of antidepressants and, perhaps, of brain stimulation. Brain stimulation methods, such as electroconvulsive therapy (ECT) has been used to treat patients with severe depression and is reported to increase BDNF levels in blood. Numerous studies has demonstrated that repetitive transcranial magnetic stimulation (rTMS) as an alternative to ECT, produced the most robust antidepressant effects, and is the most widely applied treatment protocol for major depressive disorder (MDD). Theta-burst stimulation (TBS) is a novel form of rTMS, and has recently emerged as a method with the potential to produce similar anti-depressant effects much more rapidly than traditional repetitive TMS protocols. It is presumed that BDNF mediates the therapeutic benefits of brain rTMS, but previous results are contradictory.

Specific Aims:

The study is a four-week randomized, double-blind, sham-controlled study comparing pre- and post-treatment serum BDNF levels of patients with MDD, who receive active or sham of prolonged intermittent TBS (piTBS) treatment.

Method:

During the four-week double-blind phase of active or sham piTBS treatment, piTBS sessions are scheduled daily in a 5-day sequence for 10 sessions over two weeks. Symptomatic ratings and serum BDNF measurement are administered at baseline (W0, before brain stimulation), at the end of Week 2 brain stimulation treatments, and at the two-week follow-up after the treatment (Week 4). Otherwise, the symptomatic changes are also evaluated at the end of Week 1 brain stimulation. The study include sixty patients with major depression and all participants are randomly allocated (1:1) to groups receiving either active or sham piTBS group. The aim of the present study is to explore the effect of piTBS therapy on serum BDNF levels and change of depression symptom rating scale, as well as their associations in patients with MDD.

ELIGIBILITY:
Inclusion Criteria:

1. age between 20 and 65 years;
2. fulfilling the Diagnostic and Statistical Manual version 5 (DSM-5) criteria of Major depressive disorder assessed by the Structured Clinical Interview

Exclusion Criteria:

1. Inability to provide informed consent or comprehend the study procedure;
2. A major psychiatric illness including schizophrenia spectrum disorder, bipolar spectrum disorder, and major depressive disorder with psychotic features.
3. A current DSM-5 diagnosis of substance use disorder except nicotine use disorder or the use of one to two low-potency benzodiazepine tablets for sleep impairment;
4. Have known preexisting noise-induced hearing loss, concurrent treatment with ototoxic medications, or with cochlear implants.
5. Unstable medical illness, including malignancy, uncontrolled diabetes mellitus, unstable cardiac disease or recent myocardial infarction, or cerebrovascular or cardiovascular risk factors that require intensive medical management
6. On medications known to lower seizure threshold (e.g., TCA, bupropion, clozapine)
7. Implants controlled by physiological signals, including pacemaker, implantable cardioverter defibrillator, cochlear implant.
8. Metallic objects in the head, including stenting, suture.
9. Elevated risk of seizure due to traumatic brain history, seizure history, and head trauma, intracranial lesion, and alcohol or benzodiazepines withdrawal syndrome, stimulant intoxication.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in depression severity | Before intervention (week 0) and after intervention (week 2)
  Measured by Montgomery-Asberg Depression Rating Scale (MADRS)

SECONDARY OUTCOMES:
Change in brain-derived neurotrophic factor (BDNF) | Before intervention (week 0) and after intervention (week 2)
  Serum level of BDNF

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei City Hospital, Taipei, Taipei CITY, Taiwan

IPD SHARING:
Plan to Share IPD: No